CLINICAL TRIAL: NCT00830856
Title: Randomized Control Trial of Early vs Delayed ART in the Treatment of Cryptococcal Meningitis.
Brief Title: Early Versus Delayed Antiretroviral Therapy (ART) in the Treatment of Cryptococcal Meningitis in Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zimbabwe (Other)
Collaborators: AIDS Care Research in Africa (Other)
Responsible Party: Principal Investigator, Chiratidzo Ndhlovu, Associate Professor, University of Zimbabwe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZimCrypto03
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Cryptococcal Meningitis; HIV Infections
Keywords: Cryptococcal Meningitis; HIV; Fluconazole; Antiretroviral therapy; Africa; treatment naive
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections | interventions — Fluconazole; Stavudine; Lamivudine; Nevirapine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Early initiation of antiretroviral therapy. Patients in this treatment group were started on Fluconazole 800mg by mouth every day for Cryptococcal Meningitis, and within 72hrs of diagnosis were started on First line antiretroviral therapy per Zimbabwe treatment guidelines which is Stavudine, Lamivudine and Nevirapine.
  Interventions: Drug: Fluconazole; Drug: Fixed dose - Stavudine, lamivudine and Nevirapine
- 2 (Experimental): Delayed initiation of antiretroviral therapy. Patients in this treatment group were started on Fluconazole 800mg by mouth every day for Cryptococcal Meningitis, and after completion of high dose fluconazole for 10 weeks, the patients in this group were started on First line antiretroviral therapy per Zimbabwe treatment guidelines which is Stavudine, Lamivudine and Nevirapine.
  Interventions: Drug: Fluconazole; Drug: Fixed dose - Stavudine, Lamivudine, Nevirapine

INTERVENTIONS:
Drug: Fluconazole — Fluconazole 800mg po qday
Drug: Fixed dose - Stavudine, lamivudine and Nevirapine — Initiation within 72 hours of diagnosis of Cryptococcal meningitis.
  Arms: 1
Drug: Fixed dose - Stavudine, Lamivudine, Nevirapine — Delayed initiation of ART defined as 10 weeks after initiation of high dose fluconazole therapy.
  Arms: 2

SUMMARY:
Cryptococcal Meningitis continues to be one of the most devastating AIDS defining illness in sub-Saharan Africa. Despite the availability of azoles such as fluconazole for treatment, mortality remains high with some studies showing 100% mortality. The investigators designed a study to determine if timing of the initiation of antiretroviral therapy (ART) in patients with cryptococcal meningitis and HIV would improve survival. The investigators hypothesis was that early initiation of ART result in improved mortality for patients with HIV and cryptococcal meningitis.

DETAILED DESCRIPTION:
Cryptococcosis is an invasive fungal infection caused by an encapsulated yeast. Cryptococcosis in humans is almost always caused by Cryptococcus neoformans. The advent of the HIV epidemic has lead to a profound increase in the number of reported cases of cryptococcal meningoencephalitis throughout the world, particularly in sub-Saharan Africa. In Zimbabwe an analysis of the case reports at one of the major tertiary care hospitals showed an increase in the admission rate from meningitis between 1985-1995 from 78 to 523 cases per 100000 admissions with an increase in the number of those cases due to cryptococcosis from 5% to 46.2%.

Cryptococcosis typically develops at a CD4 count of less than 50 cells/ mm3, and is the initial AIDS defining illness in up to 50-60% of patients.

Prior to the introduction of amphotericin B, flucytosine and azoles, mortality from C neoformans meningoencephalitis was close to 100%. The introduction of amphotericin B led to a significant decrease in mortality with 60-70% of patients being successfully treated. The introduction of fluconazole prophylaxis in the 1990s lead to a significant decrease in the incidence of cryptococcosis. The use of antiretroviral therapy has also caused a significant decrease in the incidence of cryptococcal meningitis.

Due to the prohibitive cost of amphotericin B and flucytosine, in many developing countries such as Zimbabwe, the mainstay of the treatment of CM is fluconazole. The current standard treatment is with fluconazole 400mg/day for 8-10 weeks, may be too low to result in adequate CNS concentration of the drug to achieve adequate killing of C. neoformans. Clinically some physicians in Zimbabwe have noted that patients are not responding adequately to this regimen and have started to treat patients with higher doses of fluconazole. Previous studies have shown that higher doses of fluconazole can be used for the treatment of CM and are well tolerated. In our proposed study, patients will be treated with high dose oral fluconazole at 800mg/day for a total 10 week period.

The advent of the increased access to ART in sub-Saharan Africa provides an additional opportunity to improve morbidity and mortality in all AIDS patients. There are as yet no definitive studies to indicate if there is an advantage to immediate ART therapy in the setting of acute CM compared to deferring therapy after the first 10 weeks of intensive CM therapy. This study is designed to address this question and provide physicians in sub-Saharan Africa with evidence based guidelines for the appropriate management of HIV positive patients with acute presentation of CM.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection documented by a positive HIV antibody test at enrollment;
* Adult men and women (age>18);
* Cryptococcal meningitis infection documented by a positive CSF CRAG or CSF identification of C. neoformans.
* Place of residence is located within a 50km radius of Harare.

Exclusion Criteria:

* Previous diagnosis (>1 week) of and treatment for cryptococcal meningitis
* Currently on ARVs, or have been intermittently on and off ART in the past.
* Concurrent use of medications that affect the metabolism of fluconazole e.g., antiseizure medications, oral hypoglycaemic agents.
* History of cardiac failure and or predisposition to arrhythmias will be excluded.
* They are pregnant or active lactation women
* History of active hepatitis or hepatic or renal dysfunction will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chiratidzo E Ndhlovu, MBChB, FRCP, Principal Investigator — University of Zimbabwe, Department of Medicine; Azure T Makadzange, MD, DPhil, Principal Investigator — University of Zimbabwe, Department of Immunology; James Hakim, MBChB, FRCP, Study Chair — University of Zimbabwe, Department of Medicine
Locations (1):
- University of Zimbabwe, College of Health Sciences, Harare, Harare, Zimbabwe

REFERENCES:
- [Derived] Makadzange AT, Ndhlovu CE, Takarinda K, Reid M, Kurangwa M, Gona P, Hakim JG. Early versus delayed initiation of antiretroviral therapy for concurrent HIV infection and cryptococcal meningitis in sub-saharan Africa. Clin Infect Dis. 2010 Jun 1;50(11):1532-8. doi: 10.1086/652652. PMID 20415574